CLINICAL TRIAL: NCT01345695
Title: Bihar Evaluation of Social Franchising and Telemedicine in India
Brief Title: Bihar Evaluation of Social Franchising and Telemedicine
Acronym: BEST
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Stanford University (Other); University College, London (Other); Sambodhi Research and Communication Pvt., Ltd. (Unknown); Public Health Foundation of India (PHFI) (Unknown); Institute of Socio-Economic Research in Development and Democracy (ISERDD) (Unknown)
Responsible Party: Sponsor
Other Study IDs: Pro00027527
Record Dates: First submitted 2011-04-25; First posted 2011-05-02 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-12

CONDITIONS: Diarrhea, Infantile; Childhood Pneumonia
Keywords: Childhood diarrhea; childhood pneumonia; telemedicine; cluster; treatment-control trial
MeSH Terms: conditions — Diarrhea, Infantile

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Treatment: Data collected on persons living in the catchment area for a WHP telemedicine center
- Control: Data collected on persons living in the catchment area where there is not a WHP telemedicine center

SUMMARY:
This study will conduct an evaluation of the World Health Partners (WHP) private provider project to see if the social franchising and telemedicine project has an impact on health outcomes in treatment vs. control areas. The evaluation will also estimate specific parameters of the WHP program that can be used to maximize financial sustainability and replicability/scalability of the program.

DETAILED DESCRIPTION:
In 2011, World Health Partners (WHP) will launch a large social franchising program of healthcare delivery in Bihar, India, with funding from the Bill and Melinda Gates Foundation (BMGF). The WHP project is particularly innovative in integrating a social franchising delivery model with a telemedicine platform. Although social franchising models of delivery are becoming increasingly common, to our knowledge, none of these efforts has been rigorously evaluated.

COHESIVE-India plans to undertake an evaluation of the BMGF-financed WHP project. The overarching focus of the evaluation project (called Bihar Evaluation of Social Franchising and Telemedicine (BEST)) is to provide evidence on the performance and effectiveness of the WHP program. In addition to studying the overall impact and effectiveness of the social franchising and telemedicine program, the evaluation will estimate how the WHP model influences outcomes related to two target diseases of interest to BMGF: childhood diarrhea and childhood pneumonia.

The Evaluation Design The core objective of the evaluation is to estimate the causal impact of the WHP program on BMGF target disease outcomes as well as other indicators of its primary health care success. The key design feature of the evaluation is that it relies on the franchisee network model of the WHP program. The evaluation design involves identifying villages in Bihar that have asymmetric digital subscriber line (ADSL) connectivity where WHP is likely to find providers who would participate in the program. The areas surrounding these villages that form catchment areas for providers will be identified; 360 such areas will be randomly sampled from the list and divided into 180 treatment and 180 control areas for implementation of the WHP program.

The study also includes a detailed costing component to estimate the costs associated with the target diseases and the benefits from the program intervention. In doing so, the evaluation strategy addresses specific policy-relevant questions about sustainability, affordability, replicability, and future Government support for privately provided healthcare options in Bihar as well as in other parts of India.

In addition, COHESIVE-India, with funding from external sources also plans to conduct studies that will provide insights on how to improve the effectiveness of the WHP model, as well as its financial sustainability. These studies include the distribution of vouchers for WHP services to estimate household's willingness to pay for them, as well experiments on financial incentives to learn how to improve the performance of network providers.

This evaluation is closely aligned with the objectives of the Government of Bihar to reduce the burden of disease. Through a rigorous evaluation of the WHP program, this study will provide evidence on whether this model of rural health service delivery is efficient and whether it can be scaled up. The stated goals of the WHP program indicate the many potential health and economic benefits to the people of Bihar. The evaluation will provide an empirical and objective assessment of the impact of WHP's effort on quality of care available in rural areas (the program anticipates a significant improvement), increases in access to healthcare providers and improved drug supply, reductions in time lapse between onset of disease and optimal care, as well as reductions in unnecessary healthcare expenditures.

ELIGIBILITY:
Inclusion Criteria:

* Households with children age < 60 months
* Persons with tuberculosis or visceral leishmaniasis
* Rural private sector medical providers

Exclusion Criteria:

* Households without children
* Households with children aged > 60 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Randomly selected residents of 12 districts in Bihar State, India.
Sampling Method: Probability Sample
Enrollment: 106380 (Estimated)
Dates: Start 2011-05; Primary Completion 2014-12 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Improvements in population based health outcomes | Baseline; 3 years
  Improvements in population based health outcomes in the treatment vs. the control areas

SECONDARY OUTCOMES:
Improvements in population based health outcomes for childhood diarrhea | Baseline; 3 years
  Proportion of children with diarrhea in the last two weeks who were treated with zinc
Improvements in population based health outcomes for childhood pneumonia | Baseline; 3 years
  Proportion of children with suspected pneumonia in the past two weeks who received a full course of antibiotics (five days)
Cost-effectiveness of the service model | Baseline; 3 years
  Through micro-experiments, we hope to gain insights on how to improve the cost effectiveness of the WHP model, as well as evaluate its financial sustainability. We will also evaluate whether the are overall improvements in the population level health indicators in the treatment vs. the control areas.

CONTACTS AND LOCATIONS:
Overall Officials: Manoj Mohanan, PhD, MPH, Principal Investigator — Duke University
Locations (1):
- BEST, Patna, Bihar, India